CLINICAL TRIAL: NCT04392895
Title: Assesment of Paraaortic Lymphadenectomy in Locally Advanced Cervical Cancer, When no Pathologic Pelvic Lymph Node on PET/CT: Retrospective Study.
Brief Title: Para Aortic Lymphadenectomy : Always ?
Acronym: PALA
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0296
Record Dates: First submitted 2020-05-13; First posted 2020-05-19 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Cervical Cancer
Keywords: Locally advanced cervical cancer, more than IB3 stage FIGO 2018; Para aortic lymphadenectomy; Laparoscopy; PET/CT
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with locally advanced cervical cancer: Patients with locally advanced cervical cancer, who had undergone a PAL
  Interventions: Procedure: Para Aortic Lymphadenectomy (PAL) by laparoscopy

INTERVENTIONS:
Procedure: Para Aortic Lymphadenectomy (PAL) by laparoscopy — Para Aortic Lymphadenectomy (PAL) by laparoscopy

SUMMARY:
Cervical cancer affects more than 3000 new cases per year in France. The treatment of stage IB3 to IVA cervical cancer is based on concomitant radio-chemotherapy. The irradiation volumes are based, according to current recommendations, on imaging examinations and / or on the results of a laparoscopic Para-aortic lymphadenectomy (PAL). There is some risk of false negatif with the PET/CT. For this reason, most of the time, PAL is offered when there is no pathological paraaortic lymph node on PET/CT. The investigators suppose that this staging surgery could be avoid when no pathological pelvic nodes are identified on PET/CT. The investigators use a retrospective study, to analyse histological report of systematic PAL, comparing to results of pre-operative PET/CT.

ELIGIBILITY:
Inclusion criteria:

- Patients with :

* locally advanced cervical cancer,
* who undergone PAL
* with pre operative PET CT, between January 2015 and december 2019

Exclusion criteria:

- patients aged under 18

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with locally advanced cervical cancer, who had undergone a PAL after a negative paraaortic PET CT, between January 2015 and december 2019
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-05-29 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
negative predictive value of PET/CT on para aortic nodes when no pathological pelvic nodes. | 1 day
  negative predictive value of PET/CT on para aortic nodes when no pathological pelvic nodes.
  The intraoperative 3D optical scan gives the tumor localization obtained by radioguided occult lesion localization thanks to pen marking left by the surgeon. The comparison is done by superimposing both acquisitions.

SECONDARY OUTCOMES:
morbidity of PAL | 1 day
  morbidity of PAL

CONTACTS AND LOCATIONS:
Overall Officials: Martha DURAES, Md, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC